CLINICAL TRIAL: NCT03340415
Title: Randomised Controlled Trial of the Timing of Full Weight Bearing Walking After Soft Tissue Hallux Valgus Surgery
Brief Title: Timing of Weight Bearing After Hallux Valgus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North District Hospital (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Orthopaedic Surgeon, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVrehab
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hallux Valgus and Bunion
Keywords: Hallux Valgus; Bunion; Post-operative; Rehabilitation; Weight Bearing Status
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Surgeon blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Rehab (No Intervention): Follow existing rehabilitation protocol of Non-weight bearing walking for 6 weeks followed by heel walking for 6 weeks; then the resumption of normal full weight-bearing walking in normal shoes at 12 weeks post-operation
- Accelerated Rehab (Experimental): Accelerated rehabilitation protocol of non-weight bearing walking for 2 weeks followed by heel walking for 10 weeks; then the resumption of normal full weight-bearing walking in normal shoes at 12 weeks post-operation
  Interventions: Other: Accelerated Rehabilitation plan

INTERVENTIONS:
Other: Accelerated Rehabilitation plan — early weight bearing after surgery
  Arms: Accelerated Rehab

SUMMARY:
Investigate the optimal timing for weight bearing after Hallux Valgus surgery. Hypothesis: Early weight bearing does not affect outcome after the Endoscopic Distal Soft Tissue Procedure for Hallux Valgus Correction.

DETAILED DESCRIPTION:
Introduction:

* Rehabilitation plans after hallux valgus/bunion surgery is varied
* From a patient's perspective, full weight bearing is paramount for quality of life and return to work/study
* No high-level study showing the optimal time to resume full weight bearing available

Hypothesis:

Early weight bearing (at 2 weeks post-op) does not affect outcome after the Endoscopic Distal Soft Tissue Procedure for Hallux Valgus correction

Trial Design:

* Parallel group
* Random allocation
* Operating Surgeon blind to randomisation

Study Setting:

* General Regional Hospital
* Single Centre

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing the EDSTP recruited

Exclusion Criteria:

* Cases requiring additional procedures (eg 2nd toe correction)
* Mental incapacitation
* Physical disability hindering rehabilitation (eg CVA, neurological disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel KK Ling, MBChB, Principal Investigator — Dept of Orthopaedics & Traumatology, the Chinese University of Hong Kong
Locations (1):
- North District Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lui TH, Ling SK, Yuen SC. Endoscopic-assisted Correction of Hallux Valgus Deformity. Sports Med Arthrosc Rev. 2016 Mar;24(1):e8-13. doi: 10.1097/JSA.0000000000000078. PMID 26752780
- [Result] Lui TH. Correction of Recurred Hallux Valgus Deformity by Endoscopic Distal Soft Tissue Procedure. Arthrosc Tech. 2017 Apr 10;6(2):e435-e440. doi: 10.1016/j.eats.2016.10.022. eCollection 2017 Apr. PMID 28580264
- [Result] Lui TH, Ng S, Chan KB. Endoscopic distal soft tissue procedure in hallux valgus surgery. Arthroscopy. 2005 Nov;21(11):1403. doi: 10.1016/j.arthro.2005.08.015. PMID 16325100
- [Result] Lui TH, Chan KB, Chan LK. Endoscopic distal soft-tissue release in the treatment of hallux valgus: a cadaveric study. Arthroscopy. 2010 Aug;26(8):1111-6. doi: 10.1016/j.arthro.2009.12.027. PMID 20678710

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 lost to follow-up. power analysis only required 40 participants.
Period: Overall Study
Arm/Group | Control Rehab | Accelerated Rehab
Started | 29 | 24
Completed | 29 | 21
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Rehab | Accelerated Rehab | Total
Number analyzed (Participants) | 29 | 21 | 50
Age, Continuous [Median (Full Range); unit: years] | 60 [25 to 71] | 60 [25 to 71] | 60 [25 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 29 | 21 | 50

OUTCOME MEASURES:

1. Primary Outcome: Hallux Valgus Angle as a Measure of the Radiological Changes
Description: Weight bearing feet X-Ray to measure radiological parameters of hallux valgus. A larger angle represents the more severe condition.
  This is the angle between the 1st metatarsal and the proximal phalanx.
Time Frame: 0, 12, 26 weeks post-surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Rehab | Accelerated Rehab
Number analyzed (Participants) | 29 | 21
degrees
  0 week | 35.6 (7.1) | 37.4 (8.0)
  12 week | 8.8 (5.2) | 7.2 (4.8)
  26 week | 11.6 (7.6) | 10.5 (6.2)

2. Primary Outcome: Inter-metatarsal Angle as a Measure of the Radiological Changes
Description: Weight bearing feet X-Ray to measure radiological parameters of hallux valgus. A larger angle represents the more severe condition.
  This is measure using the bisecting line between the 1st metatarsal and the 2nd metatarsal.
Time Frame: 0, 12, 26 weeks post-surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Rehab | Accelerated Rehab
Number analyzed (Participants) | 29 | 21
degrees
  0 week | 14.0 (3.0) | 16.4 (3.7)
  12 week | 6.2 (1.9) | 7.2 (2.2)
  26 week | 7.7 (2.7) | 7.3 (2.4)

3. Primary Outcome: Radiological Changes (Tibial Sesamoid Position)
Description: Weight bearing feet X-Ray to measure radiological parameters of hallux valgus. 4 represents the most neutral position. bigger difference from 4 means more severe condition.
  This a score from 0-7.
Time Frame: 0, 12, 26 weeks post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Rehab | Accelerated Rehab
Number analyzed (Participants) | 29 | 21
units on a scale
  0 week | 5.55 (1.2) | 5.6 (1.1)
  12 week | 2.6 (1.2) | 3.0 (0.9)
  26 week | 2.9 (1.3) | 3.0 (1.0)

4. Secondary Outcome: Foot Function (FAOS Symptoms)
Description: Calculation of foot function using the self-reported Foot and Ankle Outcome Score (FAOS): FAOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport and Recreation), and foot and ankle-related Quality of Life (QOL). The last week is taken into consideration when answering the questionnaire. Standardized answer options are given (% Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 0, 12, 26 week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control 6-wk NWB: Control group ( 6 week NWB )
- Early 2 Week NWB: Early weight bearing group （2 week)
Arm/Group | Control 6-wk NWB | Early 2 Week NWB
Number analyzed (Participants) | 29 | 21
score on a scale
  0 week | 58.3 (26.1) | 47.5 (23.9)
  12 week | 62.1 (16.1) | 76.9 (13.6)
  26 week | 81.9 (11.8) | 80.5 (15.6)

5. Secondary Outcome: Foot Function (FAOS Pain)
Description: as for outcome 4
Time Frame: 0, 12, 26 week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control 6-wk NWB | Early 2 Week NWB
Number analyzed (Participants) | 29 | 21
score on a scale
  0 week | 44 (23.8) | 47.5 (28.8)
  12 week | 66.4 (19.3) | 78.6 (11.4)
  26 week | 82.2 (15.6) | 85.5 (12.9)

6. Secondary Outcome: Foot Function (FAOS ADL)
Description: as for outcome 4
Time Frame: 0, 12, 26 week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control 6-wk NWB | Early 2 Week NWB
Number analyzed (Participants) | 29 | 21
score on a scale
  0 week | 59.7 (29.4) | 53.0 (25.6)
  12 week | 61.4 (17.3) | 81.4 (7.6)
  26 week | 84.3 (10.6) | 86.0 (8.2)

7. Secondary Outcome: Foot Function (FAOS Sport)
Description: as for outcome 4
Time Frame: 0, 12, 26 week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control 6-wk NWB | Early 2 Week NWB
Number analyzed (Participants) | 29 | 21
score on a scale
  0 week | 52.1 (29.7) | 39.8 (26.7)
  12 week | NA (NA) — The postoperative rehabilitation program prior to 12 weeks restricts the subject from sports. Thus there is no score for the "Sporting Function" section | NA (NA) — The postoperative rehabilitation program prior to 12 weeks restricts the subject from sports. Thus there is no score for the "Sporting Function" section
  26 week | 76.7 (15.7) | 77.6 (13.7)

8. Secondary Outcome: Foot Function (FAOS QoL)
Description: as for outcome 4
Time Frame: 0, 12, 26 week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control 6-wk NWB | Early 2 Week NWB
Number analyzed (Participants) | 29 | 21
score on a scale
  0 week | 41.2 (30.2) | 31.1 (23.6)
  12 week | 49.1 (20.4) | 72.6 (20.7)
  26 week | 82.4 (11.2) | 81.4 (14.9)

ADVERSE EVENTS:
Time Frame: 1 year
Description: no adverse events were encountered
Arm/Group | Control Rehab | Accelerated Rehab
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03340415/Prot_SAP_000.pdf